CLINICAL TRIAL: NCT00077181
Title: A Phase I Study of Triapine in Combination With High Dose Ara-C (Hi-DAC) in Patients With Advanced Hematologic Malignancies
Brief Title: 3-AP and High-Dose Cytarabine in Treating Patients With Advanced Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02570; UCCRC-12806B; U01CA069852 (NIH); CDR0000349659 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-02-10; First posted 2004-02-11 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Blastic Phase Chronic Myelogenous Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Cytarabine; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

ARMS (1):
- Treatment (cytarabine and triapine) (Experimental): Patients receive high-dose cytarabine IV over 2 hours on days 1-5 and triapine IV over 2 hours on days 2-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cytarabine; Drug: triapine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as cytarabine, work in different ways to stop cancer cells from dividing so they stop growing or die. 3-AP may help cytarabine kill more cancer cells by making them more sensitive to the drug. This phase I trial is studying the side effects and best dose of 3-AP when given with high-dose cytarabine in treating patients with advanced hematologic malignancies

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of 3-AP (Triapine) administered with high-dose cytarabine in patients with advanced hematologic malignancies.

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this regimen in these patients. II. Determine the effect of treatment with 3-AP (Triapine) on intracellular levels of cytarabine in these patients.

OUTLINE: This is a dose-escalation study of 3-AP (Triapine).

Patients receive high-dose cytarabine IV over 2 hours on days 1-5 and 3-AP (Triapine) IV over 2 hours on days 2-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients in each stratum receive escalating doses of 3-AP (Triapine) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed for up to 2 years.

PROJECTED ACCRUAL: A total of 6-48 patients (3-24 per stratum) will be accrued for this study within 15-24 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following hematologic malignancies:

  * Relapsed or refractory acute myeloid leukemia (AML)
  * Relapsed or refractory acute lymphoblastic leukemia
  * Secondary AML, including AML arising from antecedent hematologic diseases, such as myelodysplastic syndromes or myeloproliferative disorders OR therapy-related AML
  * Chronic myeloid leukemia in accelerated or blast phase
* Refractory to standard therapy or no standard therapy exists
* No known brain metastases
* Performance status - CALGB 0-2
* Performance status - Karnofsky 60-100%
* No G6PD deficiency
* Bilirubin < 2.0 mg/dL (unless due to Gilbert's syndrome)
* AST and ALT < 2.5 times upper limit of normal (ULN)
* Creatinine < 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No pulmonary disease requiring oxygen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to study drugs
* No neuropathy
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* No concurrent biologic agents
* At least 72 hours since prior hydroxyurea
* At least 2 weeks since other prior chemotherapy (6 weeks for mitomycin or nitrosoureas)
* No other concurrent chemotherapy
* At least 2 weeks since prior radiotherapy
* No concurrent radiotherapy
* Recovered from all prior therapy
* At least 4 weeks since prior investigational agents
* No other concurrent investigational therapy
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-01; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
MTD defined as the dose preceding that at which greater than or equal to 2 patients experience dose-limiting toxicity assessed using NCI CTCAE version 3.0 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States